CLINICAL TRIAL: NCT03394729
Title: Effect of a Propolis-containing Tablet on the Acidity of Saliva and the Amount of Adolescent Dental Plaque Microbes: a Randomized Clinical Study
Brief Title: Effect of a Propolis Tablet on the Saliva and the Amount of Adolescent Dental Plaque Microbes
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Mariana Leonel Martins, Post-graduate Student in Pediatric Dentistry, Faculty of Dentistry, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: TabletUFRJPed
Record Dates: First submitted 2017-12-26; First posted 2018-01-09 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Dental Plaque
Keywords: Propole; Xylitol; Saliva
MeSH Terms: conditions — Dental Plaque | interventions — Xylitol

STUDY DESIGN:
Intervention Model Description: Clinical trial of prevention, cross, blind, randomized controlled with two arms in the study phase 2-3.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: In the study, the principal investigator will be blind to the order of the tablets consumed by adolescents. The propolis tablets and control tablets will have a similar appearance, taste, texture and sizes, will be coded as "A" and "B" by an independent investigator and will be delivered to participants in an opaque and closed bottle. Individuals will be instructed to consume each type of tablet (propolis and propolis) twice a day (10 a.m. and 5 p.m.) for 7 days, giving a 30 day interval between test and control. Volunteers will be followed at the beginning and end of each intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propolis tablet to limit dental biofilm (Experimental): Individuals will be instructed to consume the tablet with propolis and xilytol to control dental biofilm, twice a day (at 10am and 5pm) for 7 days, giving a 30 day interval between the test and the control tablet.
  Interventions: Drug: Propolis tablet to limit dental biofilm
- Xilytol tablet to limit dental biofilm (Active Comparator): Individuals will be instructed to consume the tablet with xilytol to control dental biofilm, twice a day (at 10am and 5pm) for 7 days, giving a 30 day interval between the test and the control tablet.
  Interventions: Drug: Xilytol tablet to limit dental biofilm

INTERVENTIONS:
Drug: Propolis tablet to limit dental biofilm — The tablets will be offered in an exact number of days of use. Collection of total stimulated saliva and dental biofilm will be performed at the beginning of the study (before tablet consumption) and 7 days after the intervention. Saliva samples from each individual will be collected in separate containers as well as the biofilm samples, both at baseline and after 7 days
  Other Names: Propolis+Xylitol tablet
  Arms: Propolis tablet to limit dental biofilm
Drug: Xilytol tablet to limit dental biofilm — The tablets will be offered in an exact number of days of use. Collection of total stimulated saliva and dental biofilm will be performed at the beginning of the study (before tablet consumption) and 7 days after the intervention. Saliva samples from each individual will be collected in separate containers as well as the biofilm samples, both at baseline and after 7 days.
  Other Names: Xylitol tablet
  Arms: Xilytol tablet to limit dental biofilm

SUMMARY:
The aim of the present study was to evaluate the effect of a xylitol containing propolis tablet on the salivary pH, total microorganisms count and soluble and insoluble extracellular polysaccharide concentration of the dental biofilm of adolescents in a randomized controlled clinical trial. In addition, evaluate the acceptability of the individuals regarding the characteristics of the tablets (appearance, taste, aroma and texture) through a questionnaire. To that end, healthy adolescents between 10 and 19 years old, without active carious lesions, who seek care at the Pediatric Dentistry Clinic of the Universidade Federal do Rio de Janeiro (UFRJ) will be randomly assigned to the two groups of the study: control group (propolis- consumers of tablets with propolis), respecting an interval of 30 days of rest between the consumption of the tablets. The study will be cross-checked and the principal investigator will be blind. The tablets will be given to the participants on an exact number of days of use and they will be instructed to consume two tablets per day for 7 uninterrupted days. After 30 days of interval, they will consume the other type of tablet with the same recommendations of the first one. The total non-stimulated saliva collection will be performed at the beginning of the study (before the consumption of the tablets) and 7 days after the intervention of each type of tablet, as well as the collection of the dental biofilm. Saliva and biofilm samples from all individuals will be identified and later analyzed in the laboratory, on the same day of collection, to measure the salivary pH, with the aid of a phmeter, and evaluation of the growth of total microorganisms (CFU / mg biofilm ), respectively. From the biofilm collected and stored in saline, concentrations of soluble and insoluble extracellular polysaccharides will also be measured by means of a spectrophotometer. Statistical tests will be used to compare the groups, with a significance level of 5%. As results, the propolis-containing tablet is expected to increase the salivary pH and decrease the number of total microorganisms in the dental biofilm.

DETAILED DESCRIPTION:
Test tablets (with xylitol and propolis) and control (xylitol only) will be offered in an exact number of days of use to be consumed orally. Collection of total non-stimulated saliva and dental biofilm will be performed at the beginning of the study (before tablet consumption) and 7 days after the intervention. Saliva samples from each individual will be collected in separate containers as well as the biofilm samples, both at baseline and after 7 days, for both types of pellets and both tests. All individuals (n=300) will use the tablet with and without propolis, respecting interval of 30 days without consumption of any other tablet or substance containing propolis and/or xylitol.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 10-19 years;
* Both genders;
* Individuals without cavitary caries lesions;
* Healthy individuals without any systemic diseases.

Exclusion Criteria:

* Individuals intolerant to some component of the propolis-containing tablet;
* Subjects undergoing antimicrobial treatment during the course of the study or for a period of 30 days prior to the study;
* Individuals who used products containing xylitol up to 30 days before the start of study or during the course of the study;
* Individuals who used products containing propolis up to 30 days before the start of the study or during the course of the study;
* Individuals with orthodontic appliances;
* Individuals who are using oral mouthwashes during the period of study;
* Individuals with a history of intraoral surgery within the last 6 months;
* Individuals who are making use of products rich in polyphenols: coffee, mate, acai, in the previous period (30 days) and during the research;
* Individuals who consume alcohol.

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2020-10-21 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
Total microorganism count of adolescents biofilm | 7 days
  Effect of xylitol tablets with and without propolis on the total microorganism count of adolescents biofilm using the scattering technique, considering the number of CFU/mg of biofilm.

SECONDARY OUTCOMES:
Concentration of soluble and insoluble extracellular polysaccharides of the biofilm of adolescents | 7 days
  Effect of xylitol tablets with and without propolis on the concentration of soluble and insoluble extracellular polysaccharides of the biofilm of adolescents by means of the phenol-sulfuric method, based on the quantitative carbohydrate
Acceptability of tablets | 7 days
  The acceptability of tablets for the appearance, flavor, aroma and texture of the tablets, by adolescents, by means of a questionnaire with a scale of sensory acceptability with 9 points for each of the criteria: 9 - I liked it extremely (loved it); 8 - I liked it very much; 7 - I liked moderately; 6 - I liked it slightly; 5 - Neither liked nor disliked; 4 - I disagree slightly; 3 - I disliked moderately; 2 - I was very displeased; 1 - I greatly disliked (I hated it). The final value of this scale corresponds to the average of the scale criteria and the higher the score, the greater the sensory acceptability of the product.

CONTACTS AND LOCATIONS:
Overall Officials: Andréa F Gonçalves, Doctorate, Study Director — Universidade Federal do Rio de Janeiro
Locations (1):
- Universidade Federal do Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tulsani SG, Chikkanarasaiah N, Siddaiah SB, Krishnamurthy NH. The effect of Propolis and Xylitol chewing gums on salivary Streptococcus mutans count: a clinical trial. Indian J Dent Res. 2014 Nov-Dec;25(6):737-41. doi: 10.4103/0970-9290.152182. PMID 25728105